CLINICAL TRIAL: NCT04476498
Title: Incidence of Peristomal Infection After Pull-PEG Compared to Pull-PEG With Gastropexy
Brief Title: Prospective Comparison of Pull-PEG and Pull-PEG With Gastropexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Georg Dultz, Senior physician, Johann Wolfgang Goethe University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: JWGUHMED1-013
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2020-09

CONDITIONS: Peristomal Infection Rate; Postinterventional Bleeding; Postinterventional Mortality Rate
Keywords: Pull-PEG; Pull-PEG with gastropexy; Peristomal infection rate
MeSH Terms: interventions — Gastropexy

STUDY DESIGN:
Intervention Model Description: This study is a randomised prospective monocentric study with a one to one allocation in two different treatment arms.
Who Masked: Participant
Masking Description: The participants don't know which arm they were allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard pull-PEG (No Intervention): Standard pull-PEG
  In this group the participants receive a conventional pull-PEG as firstly described by Ponsky and Gauderer.
- Pull-PEG with gastropexy (Active Comparator): Pull-PEG with gastropexy
  In this group the participants firstly receive a gastropexy with the Funada style gastropexy device. Afterwards a conventional pull-PEG will be inserted.
  Interventions: Procedure: Pull-PEG with Gastropexy

INTERVENTIONS:
Procedure: Pull-PEG with Gastropexy — Additionally to a conventional pull-PEG a gastropexy will be performed.
  Arms: Pull-PEG with gastropexy

SUMMARY:
The study aims to compare the conventional pull-percutaneous endoscopic gastrostomy (pull-PEG) with a pull-PEG with gastropexy suture regarding the peristomal infection rate.

DETAILED DESCRIPTION:
Pull-percutaneous endoscopic gastrostomy (Pull-PEG) is currently the standard technique for enteral nutrition in patients with swallowing disorders. Fistula and peristomal infection rates are one of the most common early complications which are caused by bacterial transmission through the oropharyngeal passage of the tube and by bacterial translocation out of the stomach into the abdominal wall. Retrospective data have shown that if pull-PEGs are attached with a gastropexy suture, the abdominal wall and stomach are fixed tightly and peristomal infection rates can be reduced significantly.

This randomised study wants to compare the peristomal infection rate of standard pull-PEGs and pull-PEGs with gastropexy suture. Peristomal infection rate is detected by classical inflammation rates including erythema, exsudates, and induration, development of pus, or focal peritonitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 and over with an indication for a PEG-insertion

Exclusion Criteria:

* ASA-classification >4
* female patients who are pregnant or breast feeding
* existing contraindications for a PEG-implantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-08-03 (Actual)

PRIMARY OUTCOMES:
Peristomal infection rate | 36 months
  Peristomal infection rate will be compared after conventional pull-PEG and pull-PEG with gastropexy. Peristomal infection is detected classical inflammation parameters (erythema, indulation, exsudate, ulcer and bleeding).
Postinterventional bleeding | 36 months
  Postinterventional bleeding after PEG insertion with and without gastropexy will be observed by clinical bleeding signs and control of laboratory parameters
Postinterventional occurrence of fistulas | 36 months
  Occurence of fistulas after PEG-insertion with and without gastropexy will be detected by clinical signs and laboratory parameters

CONTACTS AND LOCATIONS:
Overall Officials: Mireen Friedrich-Rust, Professor, Study Chair — Johann Wolfgang Goethe University Hospital
Locations (1):
- Klinikum der J. W. Goethe-Universität, Frankfurt am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No